CLINICAL TRIAL: NCT04706377
Title: Vitamin B12 Supplementation in Diabetic Neuropathy :1-year Double Blind Randomized Placebo-Controlled Trial
Brief Title: Vitamin B12 Supplementation in Diabetic Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Collaborators: University of Sheffield (Other); University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, Prof. Triantafyllos Didangelos, Associate Professor of Internal Medicine-Diabetology, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: No42439
Record Dates: First submitted 2021-01-09; First posted 2021-01-12 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Diabetes Mellitus; Diabetic Neuropathies; Diabetic Complication; Diabetic Foot
Keywords: diabetic neuropathy; vitamin B12; SUDOSCAN; metformin; diabetic foot; Diabetes Mellitus; autonomic neuropathy; peripheral neuropathy; painful neuropathy
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Neuropathies; Diabetes Complications; Diabetic Foot; Peripheral Nervous System Diseases; Neuropathy, Painful | interventions — Vitamin B 12

STUDY DESIGN:
Intervention Model Description: Double Blind Placebo Controlled Randomized Clinical Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The tablets containing B12 and placebo had a similar appearance and were packed in similar containers. Patients and health care providers did not know what each package contained.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active treatment group (Active Comparator): Patients were given oral dispersible tablet with 1000μg of vitamin B12 daily for 12 months.
  Interventions: Dietary Supplement: B12 fix 1000mcg
- Placebo group (Placebo Comparator): Patients were given placebo tablet similar to the tablet given to the active group once a day for 12 months.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: B12 fix 1000mcg — oral dispersible tablet with vitamin B12 1000mcg
  Other Names: vitamin B12
  Arms: Active treatment group
Other: Placebo — Placebo tablet
  Arms: Placebo group

SUMMARY:
This prospective double-blind placebo-controlled trial aims to investigate the safety and efficacy of oral dispersible tablet of vitamin B12 for 1 year, in 90 patients with diabetes mellitus type 2 and neuropathy.

DETAILED DESCRIPTION:
In this prospective, double-blind, placebo-controlled trial, 90 patients with type 2 diabetes on metformin treatment for at least four years, and both peripheral and autonomic diabetic neuropathy were randomized to an active treatment group (n=44) receiving B12, and a control group (n=46) receiving placebo. All patients had B12 levels less than 400 pmol/L. Subjects underwent measurement of sural nerve conduction velocity and amplitude, vibration perception threshold, and performed cardiovascular autonomic reflex tests (CARTs: Mean Circular Resultant, Valsalva test, postural index and orthostatic hypotension]). Sudomotor function was assessed with the SUDOSCAN that measures electrochemical skin conductance in hands and feet. The Michigan Neuropathy Screening Instrument Questionnaire and Examination and questionnaires to evaluate quality of life and level of pain were also used.

ELIGIBILITY:
Inclusion Criteria:

* adults (>18 years old) with Diabetes Mellitus 2
* established Diabetic neuropathy, both peripheral and autonomic (Diabetic Peripheral Neuropathy and Diabetic Autonomic Neuropathy). (Diagnosis was made with a)two or more Cardiovascular Autonomic Reflex Tests abnormal, b)abnormal nerve conduction velocity, c)abnormal Michigan Neuropathy Screening Instrument Questionnaire and Michigan Neuropathy Screening Instrument Examination ).
* good glycemic control (HbA1c between 6.5 and 7.5 %), stable in the last year before participating in the study
* metformin treatment for at least 4 years
* low vitamin B12 levels according to suggested normal values for DM2 patients over 60 years old (<400 pmol/L)

Exclusion Criteria:

* pernicious anemia,
* alcoholism
* gastrectomy
* gastric bypass surgery
* pancreatic insufficiency
* malabsorption syndromes
* chronic giardiasis
* acute infection in the last 6 months
* cardiovascular event in the last 6 months
* surgery involving small intestine or Human Immunodeficiency Virus infection.
* Patients with estimated Glomerular Filtration Rate <50 mL/min/1.73m2
* taking multivitamins or B12 supplements in the last 12 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Change in Sural Nerve Function measured by conduction velocity | 12 months
  Sural Nerve conduction velocity measured as m/s
Change in Sural Nerve Function measured by amplitude | 12 months
  Sural Nerve conduction amplitude measured as μV
Change in Michigan Neuropathy Screening Instrument Questionnaire | 12 months
  Michigan Neuropathy Screening Instrument questionnaire (The Michigan Neuropathy Screening Instrument (MNSI) includes two separate assessments, a 15-item self-administered questionnaire and a lower extremity examination. the questionnaire is scored by summing abnormal responses. Responses are added to obtain a total score. 'Yes' responses to questions 1-3, 5-6, 8-9, 11-12, 14-15 are each counted as one point. 'No' responses to questions 7 and 13 each count as one point. Question 4 was considered to be a measure of impaired circulation and question 10 a measure of general asthenia and were not included in the published scoring algorithm. A score of ≥ 7 was considered abnormal.
Change in Michigan Neuropathy Screening Instrument Examination | 12 months
  Michigan Neuropathy Screening Instrument Examination (The Michigan Neuropathy Screening Instrument (MNSI) includes two separate assessments, a 15-item self-administered questionnaire that is scored by summing abnormal responses, and a lower extremity examination that includes inspection and assessment of vibratory sensation and ankle reflexes and is scored by assigning points for abnormal findings.A score ≥ 2 was considered abnormal. Abnormality in each item is graded between 0.5 and 1 and at least more than 2 abnormal items are needed to reach the score of neuropathy. )
Change in Electrochemical Skin Conductance | 12 months
  Electrochemical Skin Conductance in hands and feet measured by SUDOSCAN
Change in Cardiovascular Autonomic Reflex Tests (CARTs) | 12 months
  CARTs were performed with Autonomic Nervous System Reader and included R-R variation during deep breathing [Mean Circular Resultant , Valsalva maneuver , 30:15 ratio expressed as postural index, and blood pressure response to standing (orthostatic hypotension)
Change in Vibration perception threshold | 12 months
  Vibration perception threshold was measured using a Biothesiometer
Change in level of pain with painDETECT questionnaire | 12 months
  painDETECT questionnaire consists of seven questions that address the quality of neuropathic pain symptoms; it is completed by the patient and no physical examination is required. The first five questions ask about the gradation of pain, scored from 0 to 5 (never = 0, hardly noticed = 1, slightly = 2; moderately = 3, strongly = 4, very strongly = 5). Question 6 asks about the pain course pattern, scored from -1 to 2, depending on which pain course pattern diagram is selected. The final score between -1 and 38, indicates the likelihood of a neuropathic pain component. A score of ≤ 12 indicates that pain is unlikely to have a neuropathic component (< 15%), while a score of ≥ 19 suggests that pain is likely to have a neuropathic component (> 90%). A score between these values indicates that the result is uncertain and a more detailed examination is required.
Change in quality of life score | 12 months
  Diabetes Quality of Life Brief Clinical Inventory (ThE DQOL questionnaire we used is a 15-items, brief-focused version of the Diabetes Quality of Life (DQOL) questionnaire developed in the DCCT and lowest score means worse quality of life whereas higher values indicate better quality of life)
serum vitamin B12 levels | 12 months
  serum vitamin B12 levels

SECONDARY OUTCOMES:
Adverse events | 12 months
  report of any adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- University General Hospital AHEPA, Thessaloniki, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No